CLINICAL TRIAL: NCT00195819
Title: A Phase 3, Multicenter Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Active Ankylosing Spondylitis
Brief Title: Safety and Efficacy of Adalimumab in Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello, Director of Clinical Project Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-606
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2010-04-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental)
  Interventions: Biological: adalimumab (D2E7)
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab (D2E7) — Adalimumab 40 mg every other week (eow)
  Other Names: ABT-D2E7; adalimumab; Humira
  Arms: Adalimumab
Biological: placebo — Placebo every other week (eow)
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and clinical efficacy of adalimumab in subjects with active ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in relatively good health (Investigator discretion) with a recent stable medical history.
* Subject met the definition of AS based on the Modified New York Criteria.
* Subject had an inadequate response to or intolerance to one or more NSAIDs as defined by the Investigator

Exclusion Criteria:

* Subject had previously received anti-TNF therapy.
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-12; Primary Completion 2004-10 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (9):
  - Site Ref # / Investigator 74, Calgary, Alberta
  - Site Ref # / Investigator 70, Edmonton, Alberta
  - Site Ref # / Investigator 79, Vancouver, British Columbia
  - Site Ref # / Investigator 64, Winnipeg, Manitoba
  - Site Ref # / Investigator 78, St. John's, Newfoundland and Labrador
  - Site Ref # / Investigator 75, Toronto, Ontario
  - Site Ref # / Investigator 63, Toronto, Ontario
  - Site Ref # / Investigator 62, Toronto, Ontario
  - Site Ref # / Investigator 77, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Revicki DA, Rentz AM, Luo MP, Wong RL. Psychometric characteristics of the short form 36 health survey and functional assessment of chronic illness Therapy-Fatigue subscale for patients with ankylosing spondylitis. Health Qual Life Outcomes. 2011 May 22;9:36. doi: 10.1186/1477-7525-9-36. PMID 21600054
- [Derived] van der Heijde D, Salonen D, Weissman BN, Landewe R, Maksymowych WP, Kupper H, Ballal S, Gibson E, Wong R; Canadian (M03-606) study group; ATLAS study group. Assessment of radiographic progression in the spines of patients with ankylosing spondylitis treated with adalimumab for up to 2 years. Arthritis Res Ther. 2009;11(4):R127. doi: 10.1186/ar2794. Epub 2009 Aug 24. PMID 19703304
- [Derived] Lambert RG, Salonen D, Rahman P, Inman RD, Wong RL, Einstein SG, Thomson GT, Beaulieu A, Choquette D, Maksymowych WP. Adalimumab significantly reduces both spinal and sacroiliac joint inflammation in patients with ankylosing spondylitis: a multicenter, randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2007 Dec;56(12):4005-14. doi: 10.1002/art.23044. PMID 18050198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The placebo group included subjects who were randomized to placebo even if they received early escape open label adalimumab. The adalimumab exposure group included subjects who were randomized to blinded adalimumab.
Groups:
- Any Adalimumab: 40 mg every other week (eow), subcutaneous (SC)
Period: Double-Blind
Arm/Group | Placebo 40 mg Every Other Week (Eow), Subcutaneous (SC) | Any Adalimumab
Started | 44 | 38
Completed | 42 | 38
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Moved | 1 | 0
Period: Open-label
Arm/Group | Placebo 40 mg Every Other Week (Eow), Subcutaneous (SC) | Any Adalimumab
Started | 0 | 82
Completed | 0 | 62
Not Completed | 0 | 20
Not completed — Adverse Event | 0 | 9
Not completed — Lack of Efficacy | 0 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Moved | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Adalimumab: By duration of exposure to any adalimumab 40 mg eow, subcutaneous
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
Age Continuous [Number; unit: participants]
  <=40 years | 35
  Between 40 and 65 years | 45
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 65
Region of Enrollment [Number; unit: participants]
  Canada | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Reduction in Signs and Symptoms as Measured by Assessments of Ankylosing Spondylitis (ASAS) 20 Response at Week 12
Description: ASAS 20 responders - improvement of >=20% and absolute improvement of >=10 units from Baseline in a visual analog scale (VAS) 0 [no disease activity]-100 [high disease activity]) for >=3 of 4 domains; Patient's Global Assessment of disease activity VAS; (0[none]-100 [severe]), Total Back Pain VAS; (0 [no pain]-100 [severe]), BAth Ankylosing Spondylitis Functional Index (BASFI) VAS (0 [easy ]-100[impossible]); and Inflammation VAS; (1 [no pain] to 10 [severe pain]) and absence of deterioration in the potential remaining domain. Applied to each scale and not to an overall global scale.
Time Frame: Week 12
Population: Full analysis set - includes all subjects who were randomized and received at least one injection of study medication. The full analysis set was analyzed by treatment group.
Measure: Number; unit: participants
Groups:
- Adalimumab; Placebo: 40 mg every other week, subcutaneous
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 38 | 44
participants
  Responder | 18 | 12
  Non-responder | 20 | 32
  Missing | 0 | 0
Statistical Analysis 1: Comparison: Adalimumab; Test type: Superiority or Other; p = 0.060, Chi-squared; Odds Ratio (OR) = 20.1, 95% CI [-0.5 to 40.7]

2. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Assessments of Ankylosing Spondylitis (ASAS) 20 - Through Week 260 of Adalimumab Exposure
Description: ASAS 20 responders - improvement of >=20% and absolute improvement of >=10 units from Baseline in a visual analog scale (VAS) 0 [no disease activity]-100 [high disease activity]) for >=3 of 4 domains; Patient's Global Assessment of disease activity VAS; (0[none]-100 [severe]), Total Back Pain VAS; (0 [no pain]-100 [severe]), BASFI VAS (0 [easy ]-100[impossible]); and Inflammation VAS; (1 [no pain] to 10 [severe pain]) and absence of deterioration in the potential remaining domain. Applied to each scale and not to an overall global scale
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: Any Adalimumab Set - includes all subjects who received at least one injection of adalimumab during the Study, in either the double-blind or the open label portion. 38 randomized to 40 mg adalimumab every other week (eow) and 44 randomized to placebo. The Any Adalimumab Set will be analyzed by duration of exposure (weeks) to adalimumab.
Measure: Number; unit: participants
Groups:
- Adalimumab: By Duration of Exposure to Adalimumab 40 mg every other week, subcutaneous
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 48
  Week 24 Responders (n=80) | 52
  Week 52 Responders (n=78) | 60
  Week 76 Responders (n=75) | 57
  Week 104 Responders (n=74) | 60
  Week 128 Responders (n=70) | 57
  Week 156 Responders (n=69) | 53
  Week 180 Responders (n=62) | 47
  Week 208 Responders (n=67) | 53
  Week 220 Responders (n=64) | 55
  Week 232 Responders (n=62) | 50
  Week 244 Responders (n=54) | 49
  Week 260 Responders (n=27) | 24

3. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured by Assessments in Ankylosing Spondylitis (ASAS) ASAS 50 Through Week 260 of Adalimumab Exposure
Description: ASAS 50 responders - improvement of >=50% and absolute improvement of >=20 units (0-100) from Baseline in visual analog scale (VAS) for >=3 of the 4 domains; Patient's Global Assessment of disease activity; (0[none]-100[severe]) VAS scale; Total Back Pain VAS; (0 [no pain]-100 [severe]); BASFI VAS; (0 [easy ]-100[impossible]) and Inflammation VAS; (1 [no pain] to 10 [severe pain]). In addition, absence of deterioration in the potential remaining domain. Applied to each scale and not overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 29
  Week 24 Responders (n=80) | 38
  Week 52 Responders (n=78) | 45
  Week 76 Responders (n=75) | 46
  Week 104 Responders (n=74) | 47
  Week 128 Responders (n=70) | 46
  Week 156 Responders (n=69) | 42
  Week 180 Responders (n=62) | 38
  Week 208 Responders (n=67) | 37
  Week 220 Responders (n=64) | 42
  Week 232 Responders (n=62) | 42
  Week 244 Responders (n=54) | 40
  Week 260 Responders (n=27) | 24

4. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Assessments of Ankylosing Spondylitis (ASAS) ASAS 70 Through Week 260 of Adalimumab Exposure
Description: ASAS 70 responders - improvement of >=70% and absolute improvement of >=30 units (0-100) from Baseline in visual analog scale (VAS) for >=3 of the 4 domains; Patient's Global Assessment of disease activity VAS; (0[none]-100[severe]) Total Back Pain VAS; (0 [no pain]-100 [severe]); BASFI VAS; (0 [easy ]-100[impossible]) and Inflammation VAS; 1 [no pain] to 10 [severe pain]). In addition, absence of deterioration in the potential remaining domain. Applied to each scale and not to an overall global scale.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 18
  Week 24 Responders (n=80) | 27
  Week 52 Responders (n=78) | 32
  Week 76 Responders (n=75) | 34
  Week 104 Responders (n=74) | 35
  Week 128 Responders (n=70) | 32
  Week 156 Responders (n=69) | 31
  Week 180 Responders (n=62) | 24
  Week 208 Responders (n=67) | 28
  Week 220 Responders (n=64) | 26
  Week 232 Responders (n=62) | 28
  Week 244 Responders (n=54) | 29
  Week 260 Responders (n=27) | 14

5. Secondary Outcome: Mean Change in Patient's Global Assessment of Disease Activity in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the effect of adalimumab 40 mg every other week (eow) on patient's global assessment of disease activity. The patient was to assess his/her disease activity in the past week using a visual analog scale (VAS) on a scale of 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.
Time Frame: Weeks 12, 24, 36, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -28.55 (26.808)
  Week 24 (n=80) | -32.43 (29.047)
  Week 52 (n=78) | -38.67 (26.255)
  Week 76 (n=75) | -40.85 (25.934)
  Week 104 (n=74) | -42.72 (24.263)
  Week 128 (n=70) | -40.99 (27.741)
  Week 156 (n=69) | -40.86 (27.203)
  Week 180 (n=62) | -41.74 (26.622)
  Week 208 (n=67) | -40.79 (26.049)
  Week 220 (n=64) | -43.41 (23.854)
  Week 232 (n=62) | -42.77 (29.574)
  Week 244 (n=54) | -51.02 (23.297)
  Week 260 (n=27) | -51.26 (18.451)

6. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Patient's Global Assessment of Disease Activity (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: The patient assesses his/her disease activity for the past week using a Patient Global Assessment of Disease on visual analog scale (VAS) with 0 being none and 100 being severe.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: Any Adalimumab Set - includes all subjects who received at least one injection of adalimumab during the Study, in either the double-blind or the open label portion. 38 randomized to 40 mmg adalimumab every other week (eow) and 44 randomized to placebo. The Any Adalimumab Set will be analyzed by duration of exposure (weeks) to adalimumab.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responder (n=82) | 53
  Week 24 Responder (n=80) | 56
  Week 52 Responder (n=78) | 61
  Week 76 Responder (n=75) | 59
  Week 104 Responder (n=74) | 64
  Week 128 Responder (n=70) | 57
  Week 156 Responder (n=69) | 57
  Week 180 Responder (n=62) | 52
  Week 208 Responder (n=67) | 56
  Week 220 Responder (n=64) | 57
  Week 232 Responder (n=62) | 53
  Week 244 Responder (n=54) | 50
  Week 260 Responder (n=27) | 26

7. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Functional Index (BASFI) in Subjects With Adalimumab Exposure Through Week 260
Description: BASFI consist of a set of 10 questions designed to determine the degree of functional limitation in subjects with AS. The BASFI score was derived based on the average of questions 1 through 10. The first 8 questions considered activities related to functional anatomy and the final 2 questions assessed the subject's ability to cope with everyday life over the last week. A 10 cm visual analog scale (VAS) was used to answer the questions and the mean of the ten scales gave the BASFI score a value between 0 (easy) and 10 (impossible).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -19.83 (23.481)
  Week 24 (n=80) | -24.39 (23.559)
  Week 52 (n=78) | -27.83 (25.325)
  Week 76 (n=75) | -30.42 (24.607)
  Week 104 (n=74) | -30.51 (23.382)
  Week 128 (n=70) | -30.67 (24.209)
  Week 156 (n=69) | -30.12 (24.437)
  Week 180 (n=62) | -28.76 (24.060)
  Week 208 (n=67) | -29.81 (23.976)
  Week 220 (n=64) | -30.47 (23.333)
  Week 232 (n=62) | -31.35 (22.964)
  Week 244 (n=54) | -36.65 (21.847)
  Week 260 (n=27) | -30.83 (22.174)

8. Secondary Outcome: BASFI (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: BASFI consisted of 10 Visual Analog Scale (VAS) questions with a response ranging from 0 (easy) to 100 (impossible). The BASFI score was derived based on the average of questions 1 through 10. A responder is a subject who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responder (n=82) | 46
  Week 24 Responder (n=80) | 52
  Week 52 Responder (n=78) | 53
  Week 76 Responder (n-75) | 55
  Week 104 Responder (n=74) | 55
  Week 128 Responder (n=70) | 51
  Week 156 Responder (n=69) | 50
  Week 180 Responder (n=62) | 45
  Week 208 Responder (n=67) | 51
  Week 220 Responder (n=64) | 47
  Week 232 Responder (n=62) | 48
  Week 244 Responder (n=54) | 46
  Week 260 Responder (n=27) | 22

9. Secondary Outcome: Mean Change in Total Back Pain Visual Analog Scale (VAS) in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the effect of 40 mg every other week (eow) adalimumab on Total Back Pain VAS. The subject was to assess his/her disease activity in the past week using a total spine VAS on a scale 0 (no pain) to 100 (severe pain).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -29.30 (26.783)
  Week 24 (n=80) | -31.89 (29.675)
  Week 52 (n=78) | -39.46 (26.658)
  Week 76 (n=75) | -40.89 (26.375)
  Week 104 (n=74) | -43.85 (24.730)
  Week 128 (n=70) | -44.07 (25.944)
  Week 156 (n=69) | -42.67 (27.257)
  Week 180 (n=62) | -41.06 (28.604)
  Week 208 (n=67) | -42.16 (27.092)
  Week 220 (n=64) | -43.77 (25.228)
  Week 232 (n=62) | -42.56 (27.844)
  Week 244 (n=54) | -50.30 (23.936)
  Week 260 (n=27) | -49.41 (27.025)

10. Secondary Outcome: Total Back Pain (an Individual Component of ASAS 20) Through Week 260 of Adalimumab Exposure
Description: A responder is a subject who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline.
Time Frame: Weeks 12, 24, 52, 76, 128, 152, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responder (n=82) | 56
  Week 24 Responder (n=80) | 57
  Week 52 Responder (n=78) | 66
  Week 76 Responder (n=75) | 62
  Week 104 Responder (n=74) | 64
  Week 128 Responder (n=70) | 62
  Week 156 Responder (n=69) | 59
  Week 180 Responder (n=62) | 50
  Week 208 Responder (n=67) | 56
  Week 220 Responder (n=64) | 59
  Week 232 Responder (n=62) | 52
  Week 244 Responder (n=54) | 53
  Week 260 Responder (n=27) | 25

11. Secondary Outcome: Mean Change in Inflammation (Mean of BASDAI Questions 5 and 6) in Subjects With Adalimumab Exposure Through Week 260
Description: The inflammation score is the mean of the two morning stiffness-related BASDAI visual analog scale (VAS) scores (items 5 and 6 of the BASDAI) of 0 (none) to 10 (very severe). A decrease in inflammation represents improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
cm
  Week 12 (n=82) | -2.79 (2.650)
  Week 24 (n=80) | -3.29 (2.882)
  Week 52 (n=78) | -3.89 (2.663)
  Week 76 (n=75) | -4.12 (2.480)
  Week 104 (n=74) | -4.50 (2.465)
  Week 128 (n=70) | -4.32 (2.512)
  Week 156 (n=69) | -4.25 (2.690)
  Week 180 (n=62) | -4.21 (2.522)
  Week 208 (n=67) | -4.22 (2.553)
  Week 220 (n=64) | -4.48 (2.442)
  Week 232 (n=62) | -4.51 (2.786)
  Week 244 (n=54) | -4.96 (2.357)
  Week 260 (n=27) | -5.21 (2.375)

12. Secondary Outcome: Inflammation (Individual Component of ASAS 20) (Mean of BASDAI Questions 5 and 6) Through Week 260 of Adalimumab Exposure
Description: A responder is a subject who demonstrates an absolute improvement of at least 10 units and a percentage improvement of at least 20% from Baseline in inflammation (mean of the BASDAI questions 5 and 6 on scale of 0 [none] to 10 [very severe].
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: particpants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
particpants
  Week 12 Responder (n=82) | 52
  Week 24 Responder (n=80) | 59
  Week 52 Responder (n=78) | 66
  Week 76 Responder (n=75) | 64
  Week 104 Responder (n=74) | 65
  Week 128 Responder (n=70) | 61
  Week 156 Responder (n=69) | 55
  Week 180 Responder (n=62) | 53
  Week 208 Responder (n=67) | 58
  Week 220 Responder (n=64) | 57
  Week 232 Responder (n=62) | 53
  Week 244 Responder (n=54) | 49
  Week 260 Responder (n=27) | 25

13. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 20 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 100(very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 (none) to 10 (very severe). Improvement in BASDAI by 20% was assessed. BASDAI Scoring:
  1. Measure each item of the BASDAI in centimeters (out of a total of 10)
  2. BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
Participants
  Week 12 Responders (n=82) | 61
  Week 24 Responders (n=80) | 61
  Week 52 Responders (n=78) | 64
  Week 76 Responders (n=75) | 64
  Week 104 Responders (n=74) | 65
  Week 128 Responders (n=70) | 60
  Week 156 Responders (n=69) | 59
  Week 180 Responders (n=62) | 55
  Week 208 Responders (n=67) | 61
  Week 220 Responders (n=64) | 58
  Week 232 Responders (n=62) | 57
  Week 244 Responders (n=54) | 51
  Week 260 Responders (n=27) | 26

14. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 100 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. Improvement in BASDAI by 50% was assessed. BASDAI Scoring:
  1. Measure each item of the BASDAI in centimeters (out of a total of 10)
  2. BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 32
  Week 24 Responders (n=80) | 41
  Week 52 Responders (n=78) | 48
  Week 76 Responders (n=75) | 52
  Week 104 Responders (n=74) | 52
  Week 128 Responders (n=70) | 45
  Week 156 Responders (n=69) | 51
  Week 180 Responders (n=62) | 43
  Week 208 Responders (n=67) | 46
  Week 220 Responders (n=64) | 48
  Week 232 Responders (n=62) | 47
  Week 244 Responders (n=54) | 42
  Week 260 Responders (n=27) | 25

15. Secondary Outcome: Number of Subjects With a Reduction of Signs and Symptoms as Measured in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 70 Through Week 260 of Adalimumab Exposure
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 100 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. Improvement in BASDAI by 70% was assessed. BASDAI Scoring:
  1. Measure each item of the BASDAI in centimeters (out of a total of 10)
  2. BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 24
  Week 24 Responders (n=80) | 32
  Week 52 Responders (n=78) | 34
  Week 76 Responders (n=75) | 37
  Week 104 Responders (n=74) | 35
  Week 128 Responders (n=70) | 37
  Week 156 Responders (n=69) | 34
  Week 180 Responders (n=62) | 28
  Week 208 Responders (n=67) | 35
  Week 220 Responders (n=64) | 31
  Week 232 Responders (n=62) | 35
  Week 244 Responders (n=54) | 30
  Week 260 Responders (n=27) | 14

16. Secondary Outcome: Mean Change in BASDAI in Subjects With Adalimumab Exposure Through Week 260
Description: The BASDAI is a questionnaire with 6 questions that subject completes by marking answers on a 10-cm Visual Analog Scale (VAS) during the last week with responses that range from 0 (none) to 100 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 (none) to 10 (severe). A decrease in BASDAI represents improvement. BASDAI Scoring: 1) Measure each item of the BASDAI in centimeters (out of a total of 10) 2) BASDAI Score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
cm
  Week 12 (n=82) | -2.48 (2.305)
  Week 24 (n=80) | -2.96 (2.694)
  Week 52 (n=78) | -3.41 (2.511)
  Week 76 (n=75) | -3.70 (2.486)
  Week 104 (n=74) | -3.83 (2.392)
  Week 128 (n=70) | -3.64 (2.536)
  Week 156 (n=69) | -3.63 (2.583)
  Week 180 (n=62) | -3.60 (2.338)
  Week 208 (n=67) | -3.70 (2.367)
  Week 220 (n=64) | -3.83 (2.384)
  Week 232 (n=62) | -3.80 (2.538)
  Week 244 (n=54) | -4.36 (2.214)
  Week 260 (n=27) | -4.48 (2.011)

17. Secondary Outcome: Mean Change in C-Reactive Protein (CRP) (mg/dL) in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the mean changes in CRP in subjects with adalimumab exposure from Baseline through 5 years. The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation via the use of an ultrasensitive assay. A decrease in the level of CRP indicate reduction in inflammation. A decrease in CRP indicates improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mg/dL
  Week 12 (n=82) | -1.81 (2.782)
  Week 24 (n=80) | -1.81 (2.824)
  Week 52 (n=78) | -1.60 (3.581)
  Week 76 (n=75) | -1.86 (2.897)
  Week 104 (n=74) | -1.90 (2.850)
  Week 128 (n=70) | -1.92 (3.028)
  Week 156 (n=69) | -1.83 (3.060)
  Week 180 (n=62) | -1.99 (2.995)
  Week 208 (n=67) | -1.89 (3.063)
  Week 220 (n=64) | -2.00 (3.117)
  Week 232 (n=62) | -1.67 (3.267)
  Week 244 (n=54) | -2.07 (3.252)
  Week 260 (n=27) | -1.27 (1.513)

18. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured in Assessments of Ankylosing Spondylitis (ASAS) 40 - Through Week 260 of Adalimumab Exposure
Description: ASAS 40 responder: improvement of >= 40% and absolute improvement of >= 20 units (on a scale of 0 to 100) in >= 3 of the 4 domains: Patient global assessment (VAS score [0-100 scale]); Pain (Total Back Pain VAS score 0-100 scale); Function (BASFI score 0-100 scale); Inflammation (the mean of the two morning stiffness-related BASDAI VAS scores (i.e. the average of items 5 and 6 of the BASDAI. Applied to each scale. In addition, absence of deterioration in the potential remaining domain, where deterioration is defined as a net worsening of > 0 units (on a scale of 0 to 100).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244 and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 34
  Week 24 Responders (n=80) | 41
  Week 52 Responders (n=78) | 48
  Week 76 Responders (n=75) | 50
  Week 104 Responders (n=74) | 52
  Week 128 Responders (n=70) | 47
  Week 156 Responders (n=69) | 45
  Week 180 Responders (n=62) | 40
  Week 208 Responders (n=67) | 44
  Week 220 Responders (n=64) | 48
  Week 232 Responders (n=62) | 45
  Week 244 Responders (n=54) | 42
  Week 260 Responders (n=27) | 22

19. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured in Assessments of Ankylosing Spondylitis Ankylosing Spondylitis (ASAS) 5/6 in Subjects With Adalimumab Exposure Through Week 260
Description: The change in ASAS 5/6 was evaluated for the effect of adalimumab on structural damage.
  ASAS 5/6 criteria is the 20% improvement in 5 out of 6 domains (physical function [BASFI], Total Back Pain, Patient's Global Assessment of Disease Activity, Inflammation [mean of Questions 5 and 6 of the BASDAI], spinal mobility [BASMI], and acute phase reactants [CRP]).
Time Frame: Weeks 12, 16, 20, 24, 30, 36, 42, 48, 52, 64, 76, 88, 104, 116, 128, 140, 156, 168, 180, 192, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 45
  Week 24 Responders (n=80) | 49
  Week 52 Responders (n=78) | 55
  Week 76 Responders (n=75) | 57
  Week 104 Responders (n=74) | 56
  Week 128 Responders (n=70) | 53
  Week 156 Responders (n=69) | 51
  Week 180 Responders (n=62) | 45
  Week 208 Responders (n=67) | 48
  Week 220 Responders (n=64) | 47
  Week 232 Responders (n=62) | 49
  Week 244 Responders (n=54) | 42
  Week 260 Responders (n=27) | 22

20. Secondary Outcome: Number of Subjects With a Disease Controlling Clinical Response From Adalimumab as Measured in Partial Remission Response in Subjects With Adalimumab Exposure Through Week 260
Description: Evaluation of the mean changes in BASDAI in subjects with adalimumab exposure from Baseline through 5 years for the effect of adalimumab on structural damage. Partial remission was calculated as follows: A value below 20 on a 0 - 100-point scale in each of the four domains of the ASAS (Patient's Global Assessment of Disease Activity, Pain, Function and Inflammation). Partial remission is also regarded as a low disease activity state.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 23
  Week 24 Responders (n=80) | 25
  Week 52 Responders (n=78) | 31
  Week 76 Responders (n=75) | 33
  Week 104 Responders (n=74) | 35
  Week 128 Responders (n=70) | 31
  Week 156 Responders (n=69) | 28
  Week 180 Responders (n=62) | 29
  Week 208 Responders (n=67) | 32
  Week 220 Responders (n=64) | 29
  Week 232 Responders (n=62) | 34
  Week 244 Responders (n=54) | 25
  Week 260 Responders (n=27) | 16

21. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Metrology Index (BASMI) in Subjects With Adalimumab Exposure Through Week 260
Description: BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. BASMI 0 = indicates mild disease involvement, 1 = moderate disease, and 2 = severe disease involvement. The results for cervical rotation and lumbar side flexion are the means of the left and right measurements. Scoring range 0-10. The higher the BASMI score, the more severe was the subject's limitation of movement due to their AS.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
cm
  Week 12 (n=82) | -0.42 (1.124)
  Week 24 (n=80) | -0.50 (1.146)
  Week 52 (n=78) | -0.61 (1.492)
  Week 76 (n=75) | -0.64 (1.321)
  Week 104 (n=74) | -0.78 (1.550)
  Week 128 (n=69) | -1.01 (1.477)
  Week (156 (n=69) | -1.00 (1.426)
  Week 180 (n=62) | -1.03 (1.746)
  Week 208 (n=67) | -1.04 (1.628)
  Week 220 (n=64) | -0.86 (1.521)
  Week 232 (n=60) | -0.88 (1.541)
  Week 244 (n=51) | -1.00 (1.659)
  Week 260 (n=27) | -0.70 (1.325)

22. Secondary Outcome: Mean Change in Edmonton Ankylosing Spondylitis Metrology Index (EDASMI) in Subjects With Adalimumab Exposure Through Week 260
Description: The EDASMI is a composite spinal mobility index comprised of 4 measures: 1) cervical rotation, 2) lumbar side flexion, 3) chest expansion, and 4) hip internal rotation spread. A grade of 0-4 scoring system was developed for each of the measures. The sum of 4 items (range 0 to 16) provide the EDASMI score. Decrease in EDASMI represents improvement. All EDASMI measures were done with a simple tape measure and recorded in centimeters (cm) by a rheumatologist and a clinician nurse.
Time Frame: Weeks 12, 24, 52, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
cm
  Week 12 (n=82) | -1.11 (1.990)
  Week 24 (n=80) | -1.16 (2.143)
  Week 52 (n=78) | -1.47 (2.408)
  Week 104 (n=75) | -1.24 (2.357)
  Week 128 (n=69) | -1.59 (3.124)
  Week 156 (n=69) | -1.50 (3.457)
  Week 180 (n=62) | -1.76 (3.227)
  Week 208 (n=67) | -1.41 (3.705)
  Week 220 (n=64) | -1.34 (3.301)
  Week 232 (n=60) | -1.65 (3.267)
  Week 244 (n=51) | -1.42 (3.199)
  Week 260 (n=27) | -1.56 (3.566)

23. Secondary Outcome: Mean Change in Chest Expansion (CE) in Subjects With Adalimumab Exposure Through Week 260
Description: The patient is in a sitting position on the examination table with the hands on the hips. A pen mark is made at the xiphisternum and a tape measure placed around the circumference of the patient's chest at this level. The patient is asked to take a deep breath and to exhale as completely as possible while looking directly ahead. The measurement (in cm) is noted. The patient is asked to inhale as deeply as possible and the measurement (in cm) is noted. The difference in the 2 measurement points (in cm) constitutes the value for CE.
  An increase in chest expansion represents improvement
Time Frame: Weeks 12, 24, 52,104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
cm
  Week 12 (n=82) | 0.47 (1.907)
  Week 24 (n=80) | 0.66 (1.717)
  Week 52 (n=78) | 0.66 (1.803)
  Week 104 (n=75) | 0.51 (1.875)
  Week 128 (n=69) | 0.60 (2.287)
  Week 156 (n=69) | 0.49 (1.881)
  Week 180 (n=62) | 0.57 (1.960)
  Week 208 (n=67) | 0.60 (2.252)
  Week 220 (n=64) | 0.46 (2.013)
  Week 232 (n=60) | 0.44 (2.082)
  Week 244 (n=51) | 0.39 (2.074)
  Week 260 (n=27) | 0.52 (2.112)

24. Secondary Outcome: Mean Change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) in Subjects With Adalimumab Exposure Through Week 260
Description: MASES is measured by scoring of entheses of 0 (no tenderness) to 3 (severe tenderness) at 13 sites on the body. The score was derived as the sum of the 13 scores divided by 3 and the total range is 0 (no tenderness) to 13 (severe tenderness).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
Units on a scale
  Week 12 (n=82) | -2.26 (5.335)
  Week 24 (n=80) | -3.26 (4.608)
  Week 52 (n=77) | -3.61 (5.573)
  Week 76 (n=59) | -3.56 (5.392)
  Week 104 (n=74) | -3.66 (5.253)
  Week 128 (n=52) | -3.52 (5.207)
  Week 156 (n=67) | -3.27 (5.224)
  Week 180 (n=50) | -3.72 (4.887)
  Week 208 (n=66) | -4.11 (5.114)
  Week 232 (n=48) | -3.81 (5.640)
  Week 260 (n=49) | -5.47 (5.393)

25. Secondary Outcome: Mean Change in the Bath Ankylosing Spondylitis Global Index (BAS-G) in Subjects With Adalimumab Exposure Through Week 260
Description: BAS-G consisted of two questions that asked the subject to indicate, on a 10 cm VAS, the effect the disease had on their well being over 1) last week, and 2) last 6 months. BAS-G was measured by two VAS scores (0 to 100 mm) to reflect the effect of Ankylosing Spondylitis on subject's well-being over the past week and over the last 6 months, respectively. The average of these two scores was reported. The mean of the two scores give a BAS-G score of 0-10.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -23.41 (20.456)
  Week 24 (n=80) | -32.78 (23.638)
  Week 52 (n=78) | -39.40 (23.975)
  Week 76 (n=75) | -42.63 (23.133)
  Week 104 (n=74) | -44.78 (22.845)
  Week 128 (n=70) | -43.28 (25.578)
  Week 156 (n=69) | -44.30 (23.826)
  Week 180 (n=62) | -45.05 (22.934)
  Week 208 (n=67) | -45.08 (22.681)
  Week 220 (n=64) | -46.73 (21.367)
  Week 232 (n=62) | -45.56 (23.453)
  Week 244 (n=54) | -53.69 (18.349)
  Week 260 (n=27) | -50.93 (18.478)

26. Secondary Outcome: Mean Change in Swollen Joint Count for 44 Joints (44 SJC) in Subjects With Adalimumab Exposure Through Week 260
Description: Change from Baseline in the swollen joint index. An assessment of 44 joints for SJC done by physical examination. Joint swelling was classified as present ("1"), absent ("0") or injected/replaced ("9"). The joints assessed were: Sternoclavicular, Acromioclavicular, Shoulder, Elbow, Wrist, Metacarpophalangeal (1-5), Thumb interphalangeal, Proximal interphalangeal (2-5, Knee, Ankle, and Metatarsophalangeal (1-5).
Time Frame: Weeks 12, 24, 36, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on scale
  Week 12 (n=82) | -0.29 (4.171)
  Week 24 (n=80) | -1.00 (4.792)
  Week 52 (n=78) | -1.45 (4.497)
  Week 76 (n=59) | -0.92 (4.427)
  Week 104 (n=51) | -0.81 (5.789)
  Week 128 (n=70) | -0.04 (2.592)
  Week 156 (n=68) | -1.26 (5.231)
  Week 180 (n=50) | -1.38 (4.453)
  Week 208 (n=66) | -1.29 (5.737)
  Week 232 (n=48) | -0.33 (2.300)
  Week 260 (n=49) | -2.37 (5.619)

27. Secondary Outcome: Mean Change From Baseline in the Tender Joint Count for 46 Joints (TJC 46) in Subjects With Adalimumab Exposure Through Week 260 of Adalimumab Exposure
Description: Assessment of 46 joints for TJC was done by physical examination. Joint tenderness was classified as present ("1"), absent ("0") or injected/replaced ("9"). The joints assessed were: Sternoclavicular, Acromioclavicular, Shoulder, Elbow, Wrist, Metacarpophalangeal (1-5), Thumb interphalangeal, Proximal interphalangeal (2-5, Knee, Ankle, and Metatarsophalangeal (1-5).
Time Frame: Weeks 12, 24, 36, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on scale
  Week 12 (n=82) | -1.66 (6.639)
  Week 24 (n=80) | -2.36 (6.582)
  Week 52 (n=78) | -3.63 (5.920)
  Week 76 (n=59) | -3.34 (7.184)
  Week 104 (n=74) | -2.78 (7.731)
  Week 128 (n=52) | -3.10 (6.307)
  Week 156 (n=68) | -2.69 (8.086)
  Week 180 (n=50) | -2.90 (7.833)
  Week 208 (n=66) | -3.48 (7.341)
  Week 232 (n=48) | -3.23 (7.197)
  Week 260 (n=49) | -5.84 (7.290)

28. Secondary Outcome: Mean Change in Physician's Global Assessment of Disease Activity in Subjects With Adalimumab Exposure Through Week 260
Description: The physician will globally assess the subject's current disease state using a VAS scale with 0 being very good and 100 being very bad.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -24.80 (24.892)
  Week 24 (n=80) | -33.46 (28.197)
  Week 52 (n=78) | -38.68 (24.745)
  Week 76 (n=75) | -38.21 (24.570)
  Week 104 (n=74) | -41.96 (23.205)
  Week 128 (n=70) | -42.26 (23.083)
  Week 156 (n=69) | -38.75 (25.728)
  Week 180 (n=62) | -42.84 (25.870)
  Week 208 (n=66) | -41.27 (26.348)
  Week 220 (n=63) | -43.92 (22.369)
  Week 232 (n=58) | -43.60 (23.357)
  Week 244 (n=50) | -52.98 (16.340)
  Week 260 (n=27) | -50.33 (19.958)

29. Secondary Outcome: Mean Change in Nocturnal Pain in Subjects With Adalimumab Exposure Through Week 260
Description: The subject was to assess his/her nocturnal pain intensity for the past week using a Nocturnal Pain Visual Analog Scale (Nocturnal Pain VAS). The range was 0 to 100 mm with no pain being indicated by 0 and worse possible pain by 100.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
mm
  Week 12 (n=82) | -25.49 (29.566)
  Week 24 (n=80) | -28.08 (31.414)
  Week 52 (n=78) | -33.88 (30.432)
  Week 76 (n=75) | -34.87 (29.715)
  Week 104 (n=74) | -37.07 (28.661)
  Week 128 (n=70) | -36.77 (29.030)
  Week 156 (n=69) | -34.91 (30.125)
  Week 180 (n=62) | -33.50 (30.180)
  Week 208 (n=67) | -34.00 (29.757)
  Week 220 (n=64) | -35.33 (28.620)
  Week 232 (n=62) | -34.11 (30.186)
  Week 244 (n=54) | -40.61 (26.873)
  Week 260 (n=27) | -33.41 (30.147)

30. Secondary Outcome: Mean Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale in Subjects With Adalimumab Exposure Through Week 260
Description: The FACIT-Fatigue scale: overall score of 13 general questions divided into four primary Quality of Life (QoL) domains: 1) Physical Well-Being, 2) Social/Family Well-Being, 3) Emotional Well-Being, and 4) Functional Well-Being. For each question subject rates his/her condition for the past week on a 5-point scale ranging from 0 (not at all) to 4 (very much). The score ranges from 0 (highest level of fatigue) to 52 with 52 being the lowest level of fatigue.
Time Frame: Baseline and at Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
unit on a scale
  Week 12 (n=74) | 9.49 (9.994)
  Week 24 (n=53) | 9.03 (11.225)
  Week 52 (n=78) | 11.48 (10.331)
  Week 76 (n=59) | 11.61 (11.171)
  Week 104 (n=74) | 12.46 (10.520)
  Week 128 (n=52) | 11.08 (11.396)
  Week 156 (n=68) | 11.62 (11.391)
  Week 180 (n=50) | 10.56 (10.011)
  Week 280 (n=66) | 11.60 (10.761)
  Week 232 (n=48) | 10.13 (11.112)
  Week 260 (n=49) | 16.17 (9.276)

31. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Physical Component Summary [PCS] Through Week 260 of Adalimumab Exposure
Description: Change from Baseline in the SF-36 Health Survey Index completed by Subject to help subject keep track of how he/she was feeling and how well he/she was able to do usual activities. Components of the SF-36 included the PCS and MCS, respectively. An increase in SF-36 PCS or MCS indicate improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on scale
  Week 12 (n=74) | 7.60 (8.320)
  Week 24 (n=53) | 9.26 (9.389)
  Week 52 (n=78) | 10.63 (8.982)
  Week 76 (n=59) | 11.26 (8.685)
  Week 104 (n=74) | 11.29 (9.668)
  Week 128 (n=50) | 11.76 (8.868)
  Week 156 (n=68) | 11.73 (9.726)
  Week 180 (n=48) | 10.74 (10.781)
  Week 208 (n=60) | 12.42 (9.925)
  Week 232 (n=21) | 10.88 (10.401)
  Week 260 (n=5) | 12.19 (8.410)

32. Secondary Outcome: Number of Subjects With SF-36 Physical Component Summary (PCS) of Minimal Clinically Important Difference (MCID) Response Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0(no functioning)to 100 (highest level of functioning).
  Responders were subjects with MCID > 3 points. Minimal clinically important difference (MCID) for PCS was determined by a >= 3.0 point increase during exposure to adalimumab.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=74) | 51
  Week 24 Responders (n=53) | 41
  Week 52 Responders (n=78) | 65
  Week 76 Responders (n=59) | 50
  Week 104 Responders (n=74) | 61
  Week 128 Responders (n=50) | 43
  Week 156 Responders (n=68) | 56
  Week 180 Responders (n=48) | 38
  Week 208 Responders (n=60) | 49
  Week 232 Responders (n=21) | 15
  Week 260 Responders (n=5) | 4

33. Secondary Outcome: Mean Change in the SF-36 Health Survey Index Mental Component Summary [MCS] Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0 (no functioning) to 100 (highest level of functioning). Change from Baseline in the SF-36 Health Survey Index was completed by Subject. Components of the SF-36 included the PCS and MCS, respectively. An increase in SF-36 PCS or MCS indicated improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on scale
  Week 12 (n=74) | 6.91 (9.109)
  Week 24 (n=53) | 3.88 (10.617)
  Week 52 (n=78) | 6.14 (10.466)
  Week 76 (n=59) | 7.00 (9.469)
  Week 104 (n=74) | 6.45 (10.821)
  Week 128 (n=50) | 4.89 (11.234)
  Week 156 (n=68) | 5.76 (10.687)
  Week 180 (n=48) | 5.30 (11.434)
  Week 208 (n=60) | 6.85 (10.366)
  Week 232 (n=21) | 9.00 (11.213)
  Week 260 (n=5) | 9.40 (13.224)

34. Secondary Outcome: Number of Subjects With SF-36 Mental Component Summary (MCS) of Minimal Clinically Important Difference (MCID) Response Through Week 260 of Adalimumab Exposure
Description: SF-36 is a standardized survey completed by Subject, evaluating 8 aspects of functional health and well being; physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The score for a section is an average of the individual question scores, which are scaled 0 (no functioning) to 100 (highest level of functioning). Responders are subjects with MCID > 3 points. Minimal clinically important difference (MCID) for PCS was determined by a >= 3.0 point increase during exposure to adalimumab.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=74) | 49
  Week 24 Responders (n=53) | 29
  Week 52 Responders (n=78) | 50
  Week 76 Responders (n=59) | 39
  Week 104 Responders (n=74) | 46
  Week 128 Responders (n=50) | 30
  Week 156 Responders (n=68) | 42
  Week 180 Responders (n=48) | 27
  Week 208 Responders (n=60) | 41
  Week 232 Responders (n=21) | 16
  Week 260 Responders (n=5) | 4

35. Secondary Outcome: Mean Change in Health Utilities Index-3 (HUI-3) Through Week 260 of Adalimumab Exposure
Description: Change from baseline in Health Utility Index Mark 3 (HUI-3) was reported. The HUI-3 is a generic approach to the measurement of health status and assessment of HRQL. The HUI-3 was comprised of two complementary components. The first component was a multi-attribute health status classification system that was used to describe health status. The second component was a multi-attribute utility function that was used to value health status as measured within the corresponding multi-attribute health status classification system. An increase in the HUI-3 score represents improvement.
Time Frame: Weeks 24, 52, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on scale
  Week 24 (n=81) | 0.17 (0.234)
  Week 52 (n=62) | 0.21 (0.223)
  Week 104 (n=74) | 0.19 (0.245)
  Week 128 (n=47) | 0.19 (0.271)
  Week 156 (n=62) | 0.24 (0.254)
  Week 180 (n=49) | 0.23 (0.259)
  Week 208 (n=65) | 0.24 (0.257)
  Week 232 (n=47) | 0.18 (0.306)
  Week 260 (n=48) | 0.27 (0.249)

36. Secondary Outcome: Mean Change in the Ankylosing Spondylitis Quality of Life Questionaire (ASQoL) in Subjects Through Week 260 of Adalimumab Exposure
Description: ASQoL determined subject's quality of life and is comprised of 18 questions (yes or no) to be completed by the subject. Each statement on the ASQoL is given a score of "1" or "0." All item scores were summed to give a total score or index. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement.
Time Frame: Baseline and at Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
score on a scale
  Week 12 (n=74) | -3.90 (4.556)
  Week 24 (n=53) | -3.80 (4.993)
  Week 52 (n=78) | -5.40 (4.724)
  Week 76 (n=59) | -5.47 (4.830)
  Week 104 (n=74) | -5.55 (4.593)
  Week 128 (n=52) | -5.46 (4.741)
  Week 156 (n=68) | -5.51 (5.015)
  Week 180 (n=50) | -4.95 (5.415)
  Week 208 (n=66) | -5.80 (5.127)
  Week 232 (n=48) | -5.35 (5.538)
  Week 160 (n=49) | -7.46 (4.811)

37. Secondary Outcome: Number of Subjects With Ankylosing Spondylitis Quality of Life Questionaire (ASQoL) MCID Response (MCID <= -1.8 Points) Through Week 260 of Adalimumab Exposure
Description: ASQoL determined subject's quality of life comprised of 18 questions to be completed by the subject. Each statement on the ASQoL is given a score of "1" or "0." All item scores were summed to give a total score. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement. Responders are subjects with MCID <= -1.8 points. MCID was determined by a >= 1.8 score decrease during exposure to adalimumab.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=74) | 48
  Week 24 Responders (n=53) | 27
  Week 52 Responders (n=78) | 60
  Week 76 Responders (n=59) | 42
  Week 104 Responders (n=74) | 59
  Week 128 Responders (n=52) | 41
  Week 156 Responders (n=68) | 50
  Week 180 Responders (n=50) | 37
  Week 208 Responders (n=66) | 51
  Week 232 Responders (n=48) | 36
  Week 260 Responders (n=49) | 43

38. Secondary Outcome: Number of Subjects Achieving the Patient Acceptable Symptoms State Through Week 260 of Adalimumab Exposure
Description: Completed by subject at each visit. The MCIS was a patient reported outcome where the subjects were expected to respond (yes/no) to the following question:
  Considering all the different ways your disease is affecting you, if you would stay in this state for the next months, do you consider that your current state is satisfactory? An increase in PASS indicates improvement.
  During earlier weeks of the study PASS was measured/reported as minimal clinically important state (MCIS).
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 232, and 260
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
participants
  Week 12 Responders (n=82) | 35
  Week 24 Responders (n=80) | 44
  Week 52 Responders (n=78) | 50
  Week 76 Responders (n=75) | 50
  Week 104 Responders (n=71) | 49
  Week 128 Responders (n=51) | 35
  Week 156 Responders (n=68) | 48
  Week 180 Responders (n=48) | 32
  Week 208 Responders (n=64) | 42
  Week 232 Responders (n=47) | 34
  Week 260 Responders (n=46) | 37

39. Secondary Outcome: Mean Change From Baseline in Serum Matrix Metalloproteinase-3 (MMP-3) in Subjects Treated With Any Dose of Adalimumab Through Week 260 of Adalimumab Exposure
Description: Cartilage and bone degradation were assessed by evaluating changes in MMP-3. A decrease in MMP-3 represents improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
ng/mL
  Week 12 (n=73) | -29.06 (98.960)
  Week 24 (n=52) | -6.31 (20.115)
  Week 52 (n=78) | -24.89 (97.671)
  Week 76 (n=60) | -24.64 (102.536)
  Week 104 (n=74) | -23.05 (94.471)
  Week 128 (n=51) | -7.37 (21.704)
  Week 156 (n=66) | -33.71 (115.252)
  Week 180 (n=50) | -12.56 (36.045)
  Week 208 (n=62) | -31.37 (115.467)
  Week 220 (n=26) | -67.52 (169.992)
  Week 232 (n=36) | -9.88 (24.293)
  Week 244 (n=27) | -67.88 (168.991)
  Week 260 (n=27) | -11.60 (25.776)

40. Secondary Outcome: Mean Change From Baseline in Urine Type II Collagen C Telopeptide (CTX-II) in Subjects Treated With Any Dose of Adalimumab Through Week 260 of Adalimumab Exposure
Description: Cartilage and bone degradation were assessed by evaluating changes in CTX-II. A decrease in CTX-II represents improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mmolcr
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
ng/mmolcr
  Week 12 (n=74) | -72.27 (201.493)
  Week 24 (n=52) | -39.87 (173.995)
  Week 52 (n=75) | -51.56 (288.316)
  Week 76 (n=58) | -89.93 (324.185)
  Week 104 (n=73) | -65.04 (286.539)
  Week 128 (n=51) | -96.53 (293.026)
  Week 156 (n=64) | -125.92 (332.340)
  Week 180 (n=45) | -168.02 (368.086)
  Week 208 (n=55) | -172.18 (350.006)
  Week 220 (n=26) | -175.42 (387.357)
  Week 232 (n=35) | -113.54 (354.684)
  Week 244 (n=26) | -150.15 (383.965)
  Week 260 (n=24) | -141.42 (411.224)

41. Secondary Outcome: Mean Change From Baseline in Serum Type I Collagen N-telopeptide (NTx) in Subjects Treated With Any Dose of Adalimumab Through Week 260 of Adalimumab Exposure
Description: Cartilage degradation and bone resorption were assessed by evaluating changes in NTx. A decrease in NTx represents improvement.
Time Frame: Weeks 12, 24, 52, 76, 104, 128, 156, 180, 208, 220, 232, 244, and 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: NM BCE
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
NM BCE
  Week 12 (n=73) | 0.63 (3.890)
  Week 24 (n=53) | 0.33 (3.857)
  Week 52 (n=78) | -1.02 (4.539)
  Week 76 (n=60) | -0.05 (5.735)
  Week 104 (n=74) | -0.17 (3.891)
  Week 128 (n=50) | -1.00 (4.414)
  Week 156 (n=66) | -0.82 (3.749)
  Week 180 (n=50) | 0.52 (9.020)
  Week 208 (n=62) | -1.94 (4.182)
  Week 220 (n=26) | -3.10 (4.097)
  Week 232 (n=36) | -1.47 (3.020)
  Week 244 (n=27) | -4.59 (4.977)
  Week 260 (n=27) | -2.89 (2.903)

42. Secondary Outcome: Mean Change in Spinal Spondyloarthritis Research Consortium of Canada (S.P.A.R.C.C.) Magnetic Resonance Imaging (MRI) Index of Disease Activity Score at Weeks 12 and 52 of Adalimumab Exposure
Description: The S.P.A.R.C.C. MRI index is a tool for scoring inflammation and structural damage in both the spine and sacroiliac (SI) joints. The spinal SPARCC index score consists of 3 subscales (edema, intense edema, and deep edema). Edema was defined as the presence of increased STIR signal in each of 4 Discovertebral unit (DVU) quadrants and was assigned a score (0 = normal signal, 1 = increased signal). The scoring of edema was repeated for each of 3 consecutive sagittal slices with a maximum score of 12 per DVU (range for edema, 0-72). The total spinal SPARCC index score is 0 to 108.
Time Frame: Week 12 and Week 52
Population: Intent-to-treat (ITT) - analysis of all subjects with at least one Baseline MRI were included in the ITT population.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Adalimumab: Adalimumab every other week (eow)
- Placebo: (Week 52 - Placebo plus up to 40 weeks adalimumab)
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 38 | 44
score on a scale
  Week 12 | -9.9 (1.01) | -0.8 (0.94)
  Week 52 | -11.2 (1.08) | -13.7 (1.03)

43. Secondary Outcome: Mean Change in Sacroiliac (SI) Spondyloarthritis Research Consortium of Canada (S.P.A.R.C.C.) Magnetic Resonance Imaging (MRI) Index of Disease Activity Score at Weeks 12 and 52 of Adalimumab Exposure
Description: as for outcome 42
Time Frame: Weeks 12 and 52
Population: Intent-to-treat (ITT) - analysis of all subjects with at least one Baseline MRI were included in the ITT population.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Adalimumab Exposure: Adalimumab 40 mg every other week (eow)
- Placebo: (Week 52 - placebo plus up to 40 weeks of adalimumab)
Arm/Group | Adalimumab Exposure | Placebo
Number analyzed (Participants) | 38 | 44
score on a scale
  Week 12 | -4.1 (0.64) | -0.8 (0.60)
  Week 52 | -5.4 (0.34) | -5.5 (0.32)

44. Primary Outcome: Mean Change in the Modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) Compared Against a Historical Control Group (Outcomes in Ankylosing Spondylitis International Study [OASIS]) Using the ANCOVA Model Adjusting for Baseline mSASSS Score
Description: Radiographic progression was based on change in mSASSS scoring (comparison of the means) from double-blind Baseline visit to Week 104. The mSASSS is the sum of the lumbar and cervical spine score ( 0 [no change] to 72 [progression]), derived from scoring the anterior site of the lumbar spine (T12 to S1) and the cervical spine (C2 to T1) as either 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), 3 (bridging syndesmophyte), or N (vertebral body not evaluable). Data from NCT00195819 was compared with data from AS patients in OASIS.
Time Frame: Baseline and Week 104
Population: The OASIS cohort is a historical control group of Dutch, French, and Belgian patients with AS who have been followed up since 1996. These patients participated in a follow-up study on the natural course of AS with conventional (non-biologic) treatment.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Any Adalimumab: By duration of exposure to adalimumab 40 mg every other week, subcutaneous
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 70
score on a scale
  Adalimumab in M03-606 (N=70) | 0.5 (0.36)
  OASIS (N=169) | 0.9 (0.23)
Statistical Analysis 1: Comparison: Any Adalimumab; Test type: Superiority or Other; p = 0.387, ANCOVA; Mean Difference (Net) = -0.4, Standard Error of Mean 0.42

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through Week 260 of adalimumab exposure.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 20/82
Other Adverse Events (participants affected / at risk) | 78/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=82)
Diplopia (Eye disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bipolar disorder (Psychiatric disorders) | 1
Psychotic disorders (Psychiatric disorders) | 1
Abortion induced (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=82)
Iritis (Eye disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 13
Injection Site Reaction (General disorders) | 6
Bronchitis (Infections and infestations) | 7
Cellulitis (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 7
Influenza (Infections and infestations) | 14
Nasopharyngitis (Infections and infestations) | 38
Sinusitis (Infections and infestations) | 8
Tooth Abscess (Infections and infestations) | 9
Upper Respiratory Tract Infection (Infections and infestations) | 33
Urinary Tract Infection (Infections and infestations) | 6
Skin Laceration (Injury, poisoning and procedural complications) | 6
Tuberculin Test Positive (Investigations) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 11
Bursitis (Musculoskeletal and connective tissue disorders) | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 8
Neck Pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10
Tendonitis (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 20
Depression (Psychiatric disorders) | 5
Nephrolithiasis (Renal and urinary disorders) | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
The modified SASSS was pooled with a study (NCT00085644) similar in structure and sharing the same endpoints as this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.